CLINICAL TRIAL: NCT00696748
Title: A Randomized, Placebo-Controlled, Double-Blind, Parallel Group Study With Open-Label Follow-up to Investigate the Effect of IM Testosterone Undecanoate on Biochemical and Anthropometric Characteristics of Metabolic Syndrome in Hypogonadal Men
Brief Title: The Effect of IM Testosterone Undecanoate on Biochemical and Anthropometric Characteristics of Metabolic Syndrome in Hypogonadal Men
Acronym: NePlaM3
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Russian Academy of Medical Sciences (Other)
Responsible Party: Svetlana Kalinchenko, Russian Research Center for Endocrinology
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: U00006KO
Record Dates: First submitted 2008-06-11; First posted 2008-06-13 (Estimated); Last update posted 2008-06-13 (Estimated); Status verified 2008-06

CONDITIONS: Metabolic Syndrome; Hypogonadism
Keywords: metabolic syndrome; hypogonadism; testosterone undecanoate
MeSH Terms: conditions — Metabolic Syndrome; Hypogonadism | interventions — testosterone undecanoate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Men receiving Nebido
  Interventions: Drug: Nebido (testosterone undecanoate)
- 2 (Placebo Comparator): Men receiving Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nebido (testosterone undecanoate) — Nebido (testosterone undecanoate) intramuscular 4 ml by scheme
  Arms: 1
Drug: Placebo — Placebo 4 mL intramuscular
  Arms: 2

SUMMARY:
The objective of the study is to assess the effect of the testosterone therapy on the body composition, lipid and glucose metabolism, inflammatory markers in patients with metabolic syndrome and hypogonadism.

ELIGIBILITY:
Inclusion Criteria:

* A signed informed consent to participate in the study
* Men aged 35 to 70 with testosterone levels below 12 nmol/L or free testosterone below 225 pmol/L
* Presence of the metabolic syndrome according to the IDF definition

Exclusion Criteria:

* Patients under 35 or above 70 years.
* Participation in any clinical study within 30 days before the first injection of the drug
* Simultaneous participation in another clinical study
* Incapable subjects as well as prisoners
* Suspicion of a serious organic or mental disease according to medical history and/or clinical examination
* Prostate cancer, breast cancer or suspicion thereof
* Presence or history of hepatic tumors
* Acute or chronic hepatic disease
* Presence of renal diseases with renal failure
* Changes in biochemical or hematological laboratory values in spite of lack of clinical manifestations, in the investigator's opinion
* Suspected lack of the patient's compliance
* Hypersensitivity to the active substance

Ages: 35 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2005-10; Primary Completion 2009-01 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
waist-to-hip ratio | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Svetlana Kalinchenko, PhD, Principal Investigator — Scientific Center for Endocrinology, Russia
Locations (1):
- Scientific Centre for Endocrinology RAMS, Moscow, Russia

REFERENCES:
- [Derived] Lee H, Hwang EC, Oh CK, Lee S, Yu HS, Lim JS, Kim HW, Walsh T, Kim MH, Jung JH, Dahm P. Testosterone replacement in men with sexual dysfunction. Cochrane Database Syst Rev. 2024 Jan 15;1(1):CD013071. doi: 10.1002/14651858.CD013071.pub2. PMID 38224135
- [Derived] Kalinchenko SY, Tishova YA, Mskhalaya GJ, Gooren LJ, Giltay EJ, Saad F. Effects of testosterone supplementation on markers of the metabolic syndrome and inflammation in hypogonadal men with the metabolic syndrome: the double-blinded placebo-controlled Moscow study. Clin Endocrinol (Oxf). 2010 Nov;73(5):602-12. doi: 10.1111/j.1365-2265.2010.03845.x. PMID 20718771
- [Derived] Giltay EJ, Tishova YA, Mskhalaya GJ, Gooren LJ, Saad F, Kalinchenko SY. Effects of testosterone supplementation on depressive symptoms and sexual dysfunction in hypogonadal men with the metabolic syndrome. J Sex Med. 2010 Jul;7(7):2572-82. doi: 10.1111/j.1743-6109.2010.01859.x. Epub 2010 May 26. PMID 20524974